CLINICAL TRIAL: NCT03691350
Title: The Effects of a Standardized Research E-Cigarette on the Human Lung: A Clinical Trial With Bronchoscopic Biomarkers
Brief Title: Bronchoscopy in Determining the Effect of E-Cigarette Smoking on Biomarkers in the Lungs
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Peter Shields, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OSU-18044; NCI-2018-00283 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); U01DA045530 (NIH)
Record Dates: First submitted 2018-09-25; First posted 2018-10-01 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Cigarette Smoker; Current Every Day Smoker
MeSH Terms: interventions — Bronchoalveolar Lavage; Bronchoalveolar Lavage Fluid; Tobacco Products; Electronic Nicotine Delivery Systems; Nicotine Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group I (usual cigarette brand) (Active Comparator): Participants undergo bronchoscopy over 30-60 minutes at baseline. Participants continue to smoke their usual brand of cigarettes. Participants undergo a second bronchoscopy on day 71.
  Interventions: Procedure: Bronchoscopy with Bronchoalveolar Lavage; Drug: Cigarette; Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration
- Group II (SREC with nicotine) (Experimental): Participants undergo bronchoscopy over 30-60 minutes at baseline. After the baseline bronchoscopy, participants learn to use the SREC with nicotine for 2 weeks and switch completely to the SREC with nicotine starting day 15 for 8 weeks. Participants undergo a second bronchoscopy on day 71.
  Interventions: Procedure: Bronchoscopy with Bronchoalveolar Lavage; Other: Electronic Cigarette; Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration
- Group III (SREC without nicotine) (Experimental): Participants undergo bronchoscopy over 30-60 minutes at baseline. Beginning 1 week after bronchoscopy, participants learn to use the SREC without nicotine for 2 weeks and switch completely to the SREC without nicotine starting day 15 for 8 weeks. Participants will be offered varenicline to aid cessation. Participants undergo a second bronchoscopy on day 71.
  Interventions: Procedure: Bronchoscopy with Bronchoalveolar Lavage; Other: Electronic Cigarette; Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration
- Group IV (Nicotine Replacement Therapy [NRT]) (Experimental): Participants undergo bronchoscopy over 30-60 minutes at baseline. One week before the day 15 quit date, participants stop smoking using NRT comprising either patch, gum, or lozenge for 8 weeks. Participants undergo a second bronchoscopy on day 71.
  Interventions: Procedure: Bronchoscopy with Bronchoalveolar Lavage; Other: Laboratory Biomarker Analysis; Drug: Nicotine Replacement; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Bronchoscopy with Bronchoalveolar Lavage — Undergo bronchoscopy with bronchoalveolar lavage
  Other Names: bronchial washing; Bronchoscopy/Lavage
Drug: Cigarette — Smoke usual brand
  Arms: Group I (usual cigarette brand)
Other: Electronic Cigarette — Smoke SREC with nicotine
  Other Names: e-Cigarette; Electronic Nicotine Delivery System
  Arms: Group II (SREC with nicotine)
Other: Electronic Cigarette — Smoke SREC without nictoine
  Other Names: e-Cigarette; Electronic Nicotine Delivery System
  Arms: Group III (SREC without nicotine)
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Nicotine Replacement — Receive NRT comprising patch, gum, or lozenge
  Other Names: Nicotine Replacement Therapy; NRT
  Arms: Group IV (Nicotine Replacement Therapy [NRT])
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial studies biomarkers obtained by bronchoscopy (bronchoalveolar lavage and lung brushings) to determine the effect of smoking e-cigarettes on the lungs. Studying samples of lung cells from participants who smoke e-cigarettes may help doctors learn more about changes that occur in deoxyribonucleic acid and identify biomarkers related to cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess inflammatory changes over 10 weeks for lung and urine biomarkers in smokers who undergo serial bronchoscopy. The randomized trial includes four conditions: continued use (n=32), complete switching to the nicotine standardized research electronic cigarettes (e-cig) (SREC) (n=32), complete switching to the placebo (nicotine free) SREC (n=32), and complete switching to nicotine replacement therapy (NRT)(n=32).

OUTLINE: Participants are randomized to 1 of 4 groups.

GROUP I: Participants undergo bronchoscopy over 30-60 minutes at baseline. Participants continue to smoke their usual brand of cigarettes. Participants undergo a second bronchoscopy on day 71.

GROUP II: Participants undergo bronchoscopy over 30-60 minutes at baseline. After the baseline bronchoscopy, participants learn to use the SREC with nicotine for 2 weeks and switch completely to the SREC with nicotine for 2 weeks and switch completely to the SREC with nicotine starting day 15 for 8 weeks. Participants undergo a second bronchoscopy on day 71.

GROUP III: Participants undergo bronchoscopy over 30-60 minutes at baseline. After the baseline bronchoscopy, participants learn to use the SREC without nicotine for 2 weeks and switch completely to the SREC without nicotine starting day 15 for 8 weeks. Participants will be offered varenicline to aid cessation. Participants undergo a second bronchoscopy on day 71.

GROUP IV: Participants undergo bronchoscopy over 30-60 minutes at baseline. Beginning 1 week before the day 15 quit date, participants stop smoking using NRT comprising either patch, gum, or lozenge for 8 weeks. Participants undergo a second bronchoscopy on day 71.

After completion of study, participants are followed up at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Smokers who smoke >= 5 filtered cigarettes/day for >= 1 year
* No unstable or significant medical conditions as determined by medical history to ensure safety of the subject, to minimize the effects of poor health on biomarker measures and to maximize compliance to study procedures
* Able to read adequately to complete the survey and related study documents or give consent
* Subject has provided written informed consent to participate in the study

Exclusion Criteria:

* Regular consumption of roll your own cigarettes
* Immune system disorders requiring medication
* Prior diagnosis of chronic pulmonary disease (e.g., asthma with regular use of medications, chronic obstructive pulmonary disease [COPD], chronic bronchitis, and restrictive lung disease)
* Acute bronchitis or pneumonia within 1 year
* Reported history of diagnosed kidney or liver disease
* Any medical disorder that will increase the risk from bronchoscopy, affect biomarker data, or increase risk of an adverse effect from e-cig use
* General anesthesia within 1 year
* Regular use of inhalant medications in the last 2 months
* Use of antibiotics in prior 30 days
* Use of steroids, including corticosteroids, in prior 30 days
* Allergies to study medications, such as, lidocaine, Versed, fentanyl or Cetacaine
* Allergies to propylene glycol/glycerin or flavors
* History of hypersensitivity to varenicline
* Bronchoscopy or any other lung procedure for any reason within the previous 6 months
* Current or recent (within three months) alcohol or drug abuse problems
* Regularly smoked marijuana within the prior 3 months
* Use of an e-cigarette or other combustible tobacco products in the prior 3 months
* Currently using nicotine replacement or other tobacco cessation products (to minimize confounding effects of another product) or intention to quit in next three months
* Adverse reaction to previous e-cig use
* Body mass index (BMI) > 40 (risk of unstable airway)
* Pregnant or breastfeeding - if the subject is female, a urine pregnancy test at no cost to the subject will be done on the day of bronchoscopy
* Unable to read for comprehension or completion of study documents

Ages: 21 Years to 52 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 239 (Estimated)
Dates: Start 2018-09-17 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in cell counts and cytokines | Baseline to day 71
  Obtained via bronchoscopy with saline bronchoalveolar lavage (BAL) and bronchial brushings. Descriptive statistics and clustering (e.g., principal components analysis [PCA]), will be performed for all biomarker data measured at the different visits. Baseline data (1st bronchoscopy) will then be compared between the four groups (3 conditions and control) using a one-way analysis of variance (ANOVA). The non-parametric Kruskal-Wallis test (continuous or ordinal variables) or the chi-square test (categorical variables) will be applied when the normality assumption of the data is not met. Controls will be compared to complete substitution with the standardized research electronic cigarettes (SREC) (with and without nicotine) or nicotine replacement therapy (NRT. Generalized linear models (GLM) will be employed with measurement (cell count, gene expression, etc.) as the dependent variable, a covariable for baseline measure, and a main effect of arm.

SECONDARY OUTCOMES:
Changes in fractional exhaled nitric oxide (FeNO) levels | Baseline up to day 71
  FeNO will be measured with the NIOX VERO. Descriptive statistics and clustering (e.g. PCA), will be performed for all biomarker data measured at the different visits. Baseline data (1st bronchoscopy) will then be compared between the four groups (3 conditions and control) using a one-way ANOVA. The non-parametric Kruskal-Wallis test (continuous or ordinal variables) or the chi-square test (categorical variables) will be applied when the normality assumption of the data is not met. Controls will be compared to complete substitution with the SREC (with and without nicotine) or NRT. GLM will be employed with measurement (cell count, gene expression, etc.) as the dependent variable, a covariable for baseline measure, and a main effect of arm.
Changes in messenger (m) ribonucleic acid (RNA) and microRNA (miRNA) gene expression analyzed using sequencing | Baseline up to day 71
  Total RNA containing small RNAs will be extracted from bronchial brushing specimens using commercially available kits and used for both gene expression using the Affymetrix GeneChip Human Transcriptome Array and for miRNA expression using the Affymetrix GeneChip miRNA Array. Expression will separately be assessed through RNA sequencing. Total RNA will be extracted from lavage cells and saliva for comprehensive profiling of microbiome using commercially available kits. The ?omics? (miRNA, mRNA, and metabolomics) analysis and visualization of the data will be performed in the R statistical language. Data will be log2-transformed and normalized using either quantile normalization for gene expression (miRNA and mRNA) or normalization for metabolomics. Unsupervised clustering analysis, including PCA and hierarchical clustering will be performed to visualize natural clusters in the dataset and evaluate data quality.
Changes in deoxyribonucleic acid (DNA) gene methylation | Baseline up to day 71
  Total DNA will be extracted using commercially available kits and used for genome-wide DNA methylation profiling. Total DNA including mitochondrial DNA (mtDNA) will be extracted using commercially available kits and used for mtDNA mutation using Hiseq Next Generation Sequencing (NGS) and for mtDNA contents using quantitative polymerase chain reaction (qPCR). For preliminary identification of patterns in DNA methylation, unsupervised hierarchical clustering among the groups of samples will be performed. The Euclidian distance among the groups of samples will be calculated by the average linkage. In order to assess variance among samples, PCA will be done.
Changes in the microbiome in BAL cells and saliva | Baseline up to day 71
  Obtained via bronchoscopy with saline BAL and bronchial brushings. Samples will be analyzed to determine their bacterial composition.
Changes in untargeted metabolomics using mass spectrometry | Baseline up to day 71
  Obtained via bronchoscopy with saline BAL and bronchial brushings. The omics (miRNA, mRNA, and metabolomics) analysis and visualization of the data will be performed in the R statistical language. Data will be log2-transformed and normalized using either quantile normalization for gene expression (miRNA and mRNA) or normalization for metabolomics. Unsupervised clustering analysis, including PCA and hierarchical clustering will be performed to visualize natural clusters in the dataset and evaluate data quality.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Shields, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu